CLINICAL TRIAL: NCT01786226
Title: Treatment of Uterine Myoma With 2.5 or 5 mg Mifepristone Daily During 3 Months With 9 Months Post-treatment Follow-up. Randomized Clinical Trial.
Brief Title: Mifepristone to Treat Uterine Fibroids
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mediterranea Medica S. L. (Other)
Responsible Party: Principal Investigator, Dr. Josep LLuis Carbonell i Esteve, Medical Director, Mediterranea Medica S. L.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibroma2.5normal
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Uterine Fibroids
Keywords: leiomyoma, fibroid, mifepristone, antiprogestins
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone 2.5 mg daily for three months (Experimental): Experimental: 1
  Interventions: Drug: Oral administration of mifepristone 2.5 mg daily for three months
- Mifepristone 5 mg daily for three months (Experimental): Experimental: 2
  Interventions: Drug: Oral administration of mifepristone 5 mg daily for three months

INTERVENTIONS:
Drug: Oral administration of mifepristone 2.5 mg daily for three months — Experimental: 1
  Other Names: Low doses of antiprogestins to treat uterine fibroids
  Arms: Mifepristone 2.5 mg daily for three months
Drug: Oral administration of mifepristone 5 mg daily for three months — Experimental: 2
  Other Names: Low doses of antiprogestins to treat uterine fibroids
  Arms: Mifepristone 5 mg daily for three months

SUMMARY:
Objectives: to evaluate the efficacy, safety and quality of life by using 2.5 and mifepristone 5 mg daily doses to treat uterine fibroids over 3 months with a 9 months follow-up period.

The hypothesis of the study is that the 2.5 mg dosage resulted in a lesser reduction in fibroid size but a similar improvement in quality of life when compared to the 5 mg dose.

DETAILED DESCRIPTION:
Women, in fertile age or in premenopausal status, presenting symptomatic uterine fibroids were randomly assigned to receive 5 mg or 10 of mifepristone.

The diminishing of prevalence of symptoms attributable to uterine fibroids is the most important goal to achieve under both treatments. The possible side effects of mifepristone are slight and women's adherence to treatment is remarkable. Also the reduction of the volumes of the uterus and fibroids contribute to enhance the wellbeing of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine leiomyomata
* Reproductive age or premenopausal
* Accepting the use of non hormonal contraception
* Conformity in keeping a monthly log of all episodes of vaginal bleeding during the treatment as well as all side effects of mifepristone
* Agreeing to have ultrasound examinations in every follow-up or evaluation visit
* Agreeing to two endometrial biopsies: one before starting treatment and another in the following 10 days after treatment termination

Exclusion Criteria:

* Pregnancy or desire to become pregnant
* Breastfeeding
* Hormonal contraception or any hormonal therapy received in the last three months
* Signs or symptoms of pelvic inflammatory disease
* Adnexal masses
* Abnormal or unexplained vaginal bleeding
* Suspected or diagnosed malignant neoplastic disease
* Signs or symptoms of mental illness
* Adrenal disease
* Sickle cell anemia
* Hepatic disease
* Renal disease
* Coagulopathy
* Any other severe or important disease
* Any contraindication to receiving antiprogestins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Volume of the uterine leiomyomata with 2,5mg vs 5 mg daily of mifepristone after 3 months of treatment | 3 months
  Evaluate efficacy were the percentage changes in fibroid volumes before starting, 3 into treatment and 3, 6, and 9 months after its termination

SECONDARY OUTCOMES:
Volume of the uterus with 2,5 mg vs 5 md daily of mifepristone after 3 months of treatment. | 3 months
  Evaluate efficacy were the percentage changes in uterus volumes before starting, 3 into treatment and 3, 6, and 9 months after its termination

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Eusebio Hernández, Ciudad Habana, La Habana, Cuba

REFERENCES:
- [Result] Carbonell JL, Acosta R, Perez Y, Garces R, Sanchez C, Tomasi G. Treatment of Uterine Myoma with 2.5 or 5 mg Mifepristone Daily during 3 Months with 9 Months Posttreatment Followup: Randomized Clinical Trial. ISRN Obstet Gynecol. 2013 Jul 29;2013:649030. doi: 10.1155/2013/649030. eCollection 2013. PMID 23984082